CLINICAL TRIAL: NCT05801471
Title: An Observational Prospective Longitudinal Study for the Clinical Evaluation of Visual Field Change in Glaucoma. An Assessment of Different Models of Progression
Brief Title: Clinical Evaluation of Visual Field Change in Glaucoma: an Assessment of Different Models of Progression
Status: Recruiting | Type: Observational
Sponsor: Centervue SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: CMP_005
Record Dates: First submitted 2023-03-07; First posted 2023-04-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to collect over time a series of data in patients with glaucoma in order to evaluate different approaches in defining the progression of this pathology. These data will be collected in repeated visits over a 36-months follow-up period. At each visit, the COMPASS fundus perimeter and the Humphrey Field Analyzer (HFA) perimeter will be used to assess retinal functionality; an Optical Coherence Tomography (OCT) examination will also be performed to evaluate and obtain clinical information about the structure of the retina.

ELIGIBILITY:
Inclusion Criteria:

* Glaucomatous optic nerve head in both eyes;
* Age between 40 and 90 years;
* Best Corrected Visual Acuity ≤ 0.3 [logMar];
* Spherical refraction between -6D and +6D;
* Astigmatism between -2D and +2D.

Exclusion Criteria:

* Any ocular surgery, except for: uncomplicated cataract surgery and/or glaucoma surgery in both eyes performed within 6 months before enrollment;
* Any ocular pathology that can affect visual field other than glaucoma;
* Use of any drug that can interfere with the correct execution of perimetry or that would produce visual field loss;
* Inability to obtain reliable perimetric examinations;
* Patients with advanced glaucoma for whom, according to the clinician, a 24-2 grid is not advisable to correctly monitor the patient.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, both males and females, 40-90 years old with diagnosis of Glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2028-11-06 (Estimated); Study Completion 2028-11-06 (Estimated)

PRIMARY OUTCOMES:
Equivalence between Compass and HFA in terms of estimation of the global progression rate (MD progression slope). | 1 visit every 4 months (10 visits total), up to 3 years
  Equivalence will be defined as the 95% confidence Intervals of the mean difference between the slopes estimated with the two devices being within ± 0.1 dB/year

SECONDARY OUTCOMES:
Difference in time to identify progression between Compass and HFA using an event analysis | 1 visit every 4 months (10 visits total), up to 3 years
  Time of first detectable change [years]
Quantification of the effect of the integration of the rate of progression of structural metrics into the calculation of the rate of progression of the MD | 1 visit every 4 months (10 visits total), up to 3 years
  Quantification of the effect of the integration of the rate of progression of structural metrics (mainly the retinal nerve fiber layer thickness, microns/year) into the calculation of the rate of progression of the MD. This effect will be quantified as the improvement in the equivalence metric defined for Outcome 1
  The integration of structural OCT RNFL thickness information into progression analysis will be done using a Bayesian Linear Regression approach as suggested by Russel at al.[*]
  [*] R.A. Russel at al.; "Improved Estimates of Visual Field Progression Using Bayesian Linear Regression to Integrate Structural Information in Patients with Ocular Hypertension"; IOVS May 2012; 53(6): 2760-2769.

CONTACTS AND LOCATIONS:
Overall Officials: Luca M. Rossetti, Prof., Principal Investigator — Clinica oculistica Ospedale San Paolo
Locations (2):
- Italy (2):
  - Clinica oculistica Ospedale San Paolo, Milan, Milano
  - Glaucoma Research Center, IRCCS Fondazione "G.B. Bietti", Roma, Roma

IPD SHARING:
Plan to Share IPD: No